CLINICAL TRIAL: NCT02789839
Title: Analyses of Bone Marrow and Blood Samples From Healthy Volunteers: Focus on the redOx Metabolism - HEALTHOX
Brief Title: Analyses of Bone Marrow and Blood Samples From Healthy Volunteers: Focus on the redOx Metabolism
Acronym: HEALTHOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHAO 2016 - OH / HEALTHOX
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: redOx Metabolism
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteer (Experimental): Blood test Medullar test
  Interventions: Procedure: Blood test; Procedure: Medullar test

INTERVENTIONS:
Procedure: Blood test — Blood test of 30mL
Procedure: Medullar test — Medullar test for 2-5mL and a smear

SUMMARY:
Oxidative stress is defined by an excess of reactive oxygen species (reactive oxygen species or ROS) in cells. ROS are essential to cell life (proliferation, differentiation), including kinase activity via inhibition of phosphatases. Very low levels of ROS are observed in quiescent cells, including hematopoietic stem cells. Conversely, an excess of ROS can induce DNA damage that may lead to the destruction of the cell.

The level of ROS in cells is the result of production (mainly the NADPHoxydase and the mitochondrial respiratory chain) and their disposal via antioxidant enzymes. The hematology team of the university hospital of Tours (France) found that certain antioxidant enzymes are essential for the self-renewal of normal and leukemic cells such as glutathione peroxidase-3 (Herault O et al, J Exp Med 2012, 209:895). Their expression is modified in hematological diseases (patent WO2012085188A1 / 2012-06-28 and FR1000267310 / 2014-11-27).

Age potentially affects the level of expression of antioxidant genes, since it was established a decrease in glutathione peroxidase activity in women over 65 years (Sara E, J Gerontol A Biol Sci Med Sci 2008 63: 505). The study HEALTHOX will determine the impact of age on the oxidative metabolism of normal hematopoietic cells, and in particular the expression of antioxidant genes. It will provide a reference for analyzing disturbances of oxidative metabolism in blood diseases. The main objective is the comparison of peripheral blood and bone marrow cells depending from 3 groups of healthy volunteers: 18-39 years, 40-59 years and 60-85 years. The level of ROS and the expression of genes encoding the major antioxidant enzymes involved in the regulation of oxidative stress will be studied. The secondary objectives are to create a cell bank (blood and marrow), a blood plasma bank and a cDNA library (blood and marrow) from healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age ≥ 18 years old and ≤ 85 ans
* Informed and written consent
* Affiliation to Social Security

Exclusion Criteria:

* Subject with an history of hematologic disease
* Subject with an history of tumoral disease with chemotherapy or radiotherapy
* Subject with an history of infectious or inflammatory disease
* Subject taking a treatment in prevention of blood clots
* Subject under guardianship or protection measure
* Subject with in the last 30 days food supplement rich in antioxidant : ascorbic acid, trace elements, etc…
* Subject with in the last 30 days treatment with known effect on oxydative metabolism : N-Acetyl-Cysteine, etc…
* Participant to a drug study
* Pregnant woman

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of oxygene reactive species | 12 months
  Number of oxygene reactive species by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERAULT, PhD, Principal Investigator — CHRU TOURS
Locations (1):
- CHRU Tours, Tours, France

REFERENCES:
- [Result] Guermouche H, Ravalet N, Gallay N, Deswarte C, Foucault A, Beaud J, Rault E, Saindoy E, Lachot S, Martignoles JA, Gissot V, Suner L, Gyan E, Delhommeau F, Herault O, Hirsch P. High prevalence of clonal hematopoiesis in the blood and bone marrow of healthy volunteers. Blood Adv. 2020 Aug 11;4(15):3550-3557. doi: 10.1182/bloodadvances.2020001582. PMID 32761230